CLINICAL TRIAL: NCT01857609
Title: The Cross-Over Study to Investigate the Effect of Proton Pump Inhibitor on the Pharmacokinetics and Pharmacodynamics of Metformin in Healthy Korean Men.
Brief Title: Clinical Trial to Investigate the Effect of Proton Pump Inhibitor on the Pharmacokinetics and Pharmacodynamics of Metformin
Acronym: MPI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae Yong Chung, Assistant Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MPI
Record Dates: First submitted 2013-05-10; First posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: Metformin; Proton pump inhibitor; Drug interaction
MeSH Terms: interventions — Metformin; Pantoprazole; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metformin only (Experimental): metformin 750mg(D-1), metformin 500mg (D1)
  Interventions: Drug: Metformin
- Metformin and Pantoprazole (Experimental): pantoprazole 40mg(D-2)/ metformin 750mg + pantoprazole 40mg(D-1)/metformin 500mg + pantoprazole 40mg(D1)
  Interventions: Drug: Metformin and Pantoprazole
- Metformin and Rabeprazole (Experimental): rabeprazole 20mg(D-2)/metformin 750mg+rabeprazole 20mg(D-1)/metformin 500mg+rabeprazole 20mg(D1)
  Interventions: Drug: Metformin and Rabeprazole

INTERVENTIONS:
Drug: Metformin
  Other Names: Diabex
  Arms: Metformin only
Drug: Metformin and Pantoprazole
  Other Names: Diabex, Pantoloc
  Arms: Metformin and Pantoprazole
Drug: Metformin and Rabeprazole
  Other Names: Diabex, Pariet
  Arms: Metformin and Rabeprazole

SUMMARY:
This study aims to investigate the effect of proton pump inhibitor on the pharmacokinetics and pharmacodynamics of metformin in healthy Korean men.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subject aged 20 to 45 at screening
* A body weight in the range of 50 kg (inclusive) - 100 kg (inclusive) with ideal body weight range of +- 25%
* subjects who decide to participate voluntarily and write a informed consent form

Exclusion Criteria:

* subjects who have clinically significant disease of cardiovascular, respiratory, renal, endocrinological, hematological, gastrointestinal, neurological(central nervous system), psychiatric disorders or malignant tumor
* Subject judged not eligible for study participation by investigator.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
AUC(area under the plasma concentration-time curve) | Predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12h postdose
  AUC(area under the plasma concentration-time curve), Cmax(maximum plasma concentration), t1/2

SECONDARY OUTCOMES:
AUG(total area under the serum concentration-time curve for glucose) | predose and 15, 30, 45, 60, 90, 120, 150, 180min oral glucose tolerance test
  AUG (total area under the serum concentration-time curve for glucose) Gmax(maximum serum glucose concentration)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Yong Chung, MD, PhD, Principal Investigator — Department of Clinical Pharmacology and Therapeutics, Seoul National University Bundang Hospital, Seoul, Korea
Locations (1):
- Seoul National University Bundang Hospital, Seoul, South Korea